CLINICAL TRIAL: NCT05318885
Title: Effect of Forward-leaning Position on Vital Signs, Pain and Anxiety of Children With Acute Asthma Attacks: A Randomized Controlled Study
Brief Title: The Effect of Nebulization Positions in Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Kas Alay, Research Assistant, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0001-7140-6540
Record Dates: First submitted 2022-03-06; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Asthma Attack; Asthma in Children; Asthma Acute; Asthma
Keywords: Asthma attack; Child; Nurse; Nebulization; Chest Pain
MeSH Terms: conditions — Asthma; Chest Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Forward leaning position (Experimental): The children in asthma attacks were administered nebulization three times, during which the study group children were placed in the forward-leaning position.
  Interventions: Other: A Randomized Controlled Study
- Fowler position (No Intervention): The children in asthma attacks were administered nebulization three times, during which the control group children in the routine Fowler's position.

INTERVENTIONS:
Other: A Randomized Controlled Study — For forward-leaning position, the child is first placed on a suitable chair with a soft pillow on their knees. The child will remain in the same position for the duration of the nebulization, and the pillow provides support, ensuring the child does not get tired. The child leans forward at an angle of 45°, places their arms on the pillow as shown in the figure and holds their head upright with their eyes facing forward (slight hyperextension). The upright head position of the child prevents spillage of the liquid medicine from the nebulizer chamber.
  Arms: Forward leaning position

SUMMARY:
The purpose of this study was to establish the effect on pulse rate, oxygen saturation, respiratory rate, pain and anxiety levels of Fowler's and the forward-leaning positions during nebulization in children experiencing asthma attacks.

DETAILED DESCRIPTION:
In the first stage, data on the children who agreed to participate in the study were recorded on the "Patient Identification Form" 10 minutes before the procedure by the researcher during a face-to-face interview. The children's body temperature, oxygen saturation, pulse rate and respiratory rate were measured. Upon explaining the FPS-R, the children were asked whether they had experienced pain before treatment, and to point at the pain level felt from among the faces on the scale. Then, CSA was explained and the children, and their level of anxiety on the scale was recorded. The pre-nebulization findings were recorded.

In the second stage, the salbutamol therapy prescribed by the physician was administered to the participating children with a nebulizer three times at 20-minute intervals. During nebulization, the study group patients were placed in forward-leaning position, placing a pillow on their knees, while the control group was placed in Fowler's position on a chair. Nebulization took an average of 10 minutes for each child. Oxygen saturation, pulse and respiratory rate were recorded immediately after the mask was removed. The children were allowed to rest for 20 minutes in Fowler's position.

In the third stage, oxygen saturation, pulse and respiratory rate were determined immediately after the mask was removed following a 10-minute second nebulization. The values determined were recorded, and the children were allowed to rest for 20 minutes in Fowler's position.

In the fourth stage, oxygen saturation, pulse and respiratory rate were determined immediately after the mask was removed following the 10-minute third nebulization. The children were asked whether they had pain, and to point at the pain level represented by the faces on the scale. The patients then marked their level of anxiety on the CSA. The post-nebulization findings were recorded.

ELIGIBILITY:
Inclusion Criteria:

* To be between 6-11 ages,
* Having a body temperature below 37.2°C at admission,
* Having been prescribed nebulized salbutamol by the physician during data collection,
* Having not using bronchodilators or corticosteroid drugs within the last 6 hours,
* Having no other respiratory system disease,
* Verbal and written consent of the child and parent to participate in the study.

Exclusion Criteria:

* Administering drugs other than nebulized salbutamol to the child during data collection,
* Having an obstacle for positioning (Lordosis, kyphosis, scoliosis, chest wall deformities, previous surgical procedure, etc.),
* Child and parent not knowing Turkish.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Saturation | 90 minute
  Oxygen saturation will be monitored
Change in respiratory rate | 90 minute
  Respiratory rate will be monitored
Change in Pulse Rate | 90 minute
  Heart rate will be monitored
Change in chest pain score | 90 minute
  Pain score will be evaluated with The faces pain scale-revised (FPS-R).
Change in anxiety score | 90 minute
  Anxiety score will be evaluated with The children state anxiety scale (CSA).

CONTACTS AND LOCATIONS:
Overall Officials: Gamze KAŞ ALAY, Msc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Wilder C, Shiralkar S. Childhood asthma in the emergency department: an audit. Int Emerg Nurs. 2015 Apr;23(2):197-202. doi: 10.1016/j.ienj.2014.09.001. Epub 2014 Sep 6. PMID 25263689
- [Background] Sheldon G, Heaton PA, Palmer S, Paul SP. Nursing management of paediatric asthma in emergency departments. Emerg Nurse. 2018 Nov 6;26(4):32-42. doi: 10.7748/en.2018.e1770. Epub 2018 Oct 17. PMID 30362669
- [Background] Kocaaslan EN, Akgun Kostak M. Effect of disease management education on the quality of life and self-efficacy levels of children with asthma. J Spec Pediatr Nurs. 2019 Apr;24(2):e12241. doi: 10.1111/jspn.12241. Epub 2019 Mar 19. PMID 30887669
- [Background] Camargo CA Jr, Spooner CH, Rowe BH. Continuous versus intermittent beta-agonists in the treatment of acute asthma. Cochrane Database Syst Rev. 2003;2003(4):CD001115. doi: 10.1002/14651858.CD001115. PMID 14583926
- [Background] Iramain R, Castro-Rodriguez JA, Jara A, Cardozo L, Bogado N, Morinigo R, De Jesus R. Salbutamol and ipratropium by inhaler is superior to nebulizer in children with severe acute asthma exacerbation: Randomized clinical trial. Pediatr Pulmonol. 2019 Apr;54(4):372-377. doi: 10.1002/ppul.24244. Epub 2019 Jan 22. PMID 30672140
- [Background] Myint WW, Htay MNN, Soe HHK, Renjue L, Shirying G, Yuan NSB, et al. Effect of body positions on lungs volume in asthmatic patients: A cross-sectional study. Journal of Advances in Medical and Pharmaceutical Sciences 2017;13(4):1-6. http://doi.org/10.9734/JAMPS/2017/33901
- [Background] Ganapathi LV, Vinoth S. The estimation of pulmonary functions in various body postures in normal subjects. International Journal of Advances in Medicine 2015;2(3):250-4. https://doi.org/10.18203/2349-3933.IJAM20150554
- [Background] Martinez JA, Rodrigues HB, Portelinha AM. A novel position for postural relief of dyspnea. J Bras Pneumol. 2011 Nov-Dec;37(6):829-30. doi: 10.1590/s1806-37132011000600020. No abstract available. English, Portuguese. PMID 22241044
- [Background] Sharp JT, Drutz WS, Moisan T, Foster J, Machnach W. Postural relief of dyspnea in severe chronic obstructive pulmonary disease. Am Rev Respir Dis. 1980 Aug;122(2):201-11. doi: 10.1164/arrd.1980.122.2.201. No abstract available. PMID 7416599
- [Background] Tuncer M, Khorshtd L. Obez bireylerde pozisyonların oksijen satürasyonuna etkisi. Ege Üniversitesi Hemşirelik Fakültesi Dergisi 2018;34:54-65. https://dergipark.org.tr/tr/download/article-file/456669
- [Background] Korkmaz M, Kızılcı S. Posture and ıts effect on peripheral oxygen saturation, and some hemodynamic parameters in patients with heart failure. Turkiye Klinikleri Journal of Nursing Science 2012;4(2):85-93. https://www.turkiyeklinikleri.com/article/posture-and-its-effect-on-peripheral-oxygen-saturation-and-some-hemodynamic-parameters-in-patients-with-heart-failure-63546.html
- [Background] Baysal E, Midilli ST, Ergin E. Effects of different position changes on hemodynamic parameters and dyspnea severity in patients with dyspnea. Clinical and Experimental Health Sciences 2018;8:261-7. doi: 10.5152/clinexphealthsci.2017.751
- [Background] Mohammed J, Abdulateef A, Shittu A, Sumaila FG. Effect of different body positioning on lung function variables among patients with bronchial asthma. Archives of Physiotherapy and Global Researches 2017;21(3):7-12. http://apgr.wssp.edu.pl/wp-content/uploads/2017/12/APGR-21-3-A.pdf
- [Background] Hojat B, Mahdi E. Effect of different sitting posture on pulmonary function in students. Journal of Physiology and Pathophysiology 2011;2(2):29-33. https://academicjournals.org/article/article1381307359_Hojat%20and%20mahdi%20PDF.pdf